CLINICAL TRIAL: NCT04563468
Title: Effects of Inspiratory Muscle Training on Exertional Breathlessness in Patients With Unilateral Diaphragm Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Daniel Langer, prof. dr. PT, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S60754
Record Dates: First submitted 2020-09-09; First posted 2020-09-24 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Diaphragmatic Paralysis
Keywords: diaphragm; paralysis; dysfunction; unilateral; phrenic nerve; dyspnea
MeSH Terms: conditions — Respiratory Paralysis; Paralysis; Dyspnea

STUDY DESIGN:
Intervention Model Description: Single blind, parallel group RCT with 2:1 allocation ratio
Who Masked: Participant
Masking Description: Treatment with inspiratory muscle training will be presented to both groups of patients as active interventions (intentional deception) to increase compliance. Participants in the intervention group will be informed that they are performing a 'strength training' while participants in the control group that they are performing an 'endurance training'. Participants in the control group will be offered the active treatment upon completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength inspiratory muscle training group (Experimental): Strength IMT
  Interventions: Procedure: Strength inspiratory muscle training
- Endurance inspiratory muscle training group (Sham Comparator): Endurance IMT
  Interventions: Procedure: Endurance inspiratory muscle training

INTERVENTIONS:
Procedure: Strength inspiratory muscle training — Two training sessions per day consisting of 30 breaths (against external load of ~50% Pi,max; 4-5 minutes per session), 7 days/week (once/month supervised at the research center), for 6 months will be performed using an electronic tapered flow resistive loading (TFRL) device (POWERbreathe®KH1, HaB International Ltd., Southam, UK) according to an established method. Measurements of Pi,max will be performed every week and training loads will be increased continuously to maintain external load at ~50% of Pi,max values. Ratings of perceived inspiratory effort on a modified Borg scale (4-5 out of 10) will also be used to support decisions on increasing training load.
  Arms: Strength inspiratory muscle training group
Procedure: Endurance inspiratory muscle training — Two daily sessions of 30 breaths using TFRL device (POWERbreathe®KH1, HaB International Ltd., Southam, UK) and will train at an inspiratory load of no more than 10% of their initial Pi,max. This training load will not be changed during the entire study period. Participants in the control group will be offered the active treatment upon completion of the study.
  Arms: Endurance inspiratory muscle training group

SUMMARY:
Treatment options for unilateral diaphragm paralysis are limited. Diaphragmatic plication via mini thoracotomy is sometimes considered in the University Hospital Leuven if severe symptoms persist for longer than 12 months after initial diagnosis. Preliminary data indicate that daily inspiratory muscle strength and endurance training can lead to increased nondiaphragmatic inspiratory muscle recruitment and help those with symptoms from diaphragmatic paralysis. Randomized controlled trials comparing intervention groups with improvements achieved by natural recovery in the first months after diagnosis are however so far lacking. The objective of the current study is therefore to investigate the effects of daily inspiratory muscle training in the first 6 months following diagnosis of unilateral diaphragmatic paralysis. The investigators hypothesize that respiratory muscle training in symptomatic patients with UDP (in comparison with a control group) will reduce symptoms of exertional dyspnea (primary outcome) and will improve respiratory muscle function (at rest and during exercise) and pulmonary function (sitting and supine).

DETAILED DESCRIPTION:
1. RATIONALE AND BACKGROUND Diaphragmatic paralysis is an uncommon, yet underdiagnosed cause of dyspnea. Although the diaphragm performs most of the work, normal ventilation also requires the simultaneous contraction of other respiratory muscles (ie, scalene, parasternal portion of the internal and external intercostal muscles, sternocleidomastoid, trapezius). An increased effort in the struggle to breathe may fatigue the accessory muscles and lead to ventilatory failure. It is thus far not clear whether specific training of the respiratory muscle can improve or restore diaphragm function or accessory respiratory muscle function in these patients.

Depending on the etiology of the diaphragmatic paralysis, the prognosis of unilateral disease usually is good. Patients with phrenic injuries may recover fully or partially. At times, patients may also spontaneously recover from idiopathic disease. Patients who do not recover from unilateral diaphragmatic dysfunction generally lead relatively normal lives. Many patients however keep reporting symptoms of dyspnea that interfere with performance of daily activities. In this group, dyspnea typically develops with exertion, leading to increased ventilatory demands. Dyspnea can also be elicited by changes in posture (e.g. lying supine, bending forward). Depending on the activity profile of the subjects this might have an impact on quality of life. The investigators will therefore evaluate symptoms and recruitment of respiratory muscles of these patients during exertion (i.e. while performing an exercise test on a cycle ergometer).

The morbidity of the unilateral paralysis is mainly based on the underlying pulmonary functional status and the etiology of the paralysis. Most of the patients that are referred to the University Hospital Leuven report symptoms of dyspnea during exertion or with changes in posture. Diaphragmatic paralysis is more likely to affect the left hemidiaphragm. Unilateral diaphragmatic paralysis is characterized by abnormalities of pulmonary and respiratory muscle function. Patients develop restrictive ventilatory impairment, and the vital capacity and total lung capacity frequently are below 70% of the predicted normal values. Lung capacity is reduced further when the patient assumes the supine position.

In contrast to bilateral disease, physicians can usually diagnose unilateral paralysis with only radiographic studies. Because accessory muscle contraction may create the appearance of diaphragmatic movement, fluoroscopy studies may be misleading the physician when diagnosing bilateral diaphragmatic paralysis. In fluoroscopic sniff testing, paradoxical elevation of the paralyzed diaphragm is observed with inspiration and confirms diaphragmatic paralysis. However, the sniff test is not very specific; 6% of normal persons exhibit paradoxical motion on fluoroscopy. Computerized tomography may be indicated in certain patients to evaluate for potential causes of diaphragmatic paralysis that are due to mediastinal pathology and malignancy. MRI may be indicated in certain patients to determine the presence of pathologic conditions involving the spinal column or nerve roots that are causing diaphragmatic paralysis.

M-mode ultrasonography is a relatively simple and accurate test for diagnosing paralysis of the diaphragm in the adult population and it can be performed at the bedside. The paralyzed side shows no active caudal movement of the diaphragm with inspiration and abnormal paradoxical movement (ie, cranial movement on inspiration), particularly with the sniff test. B-mode ultrasonography of diaphragm thickness in the zone of apposition of the diaphragm to the rib cage can also provide a sensitive and specific noninvasive assessment of diaphragmatic paralysis. Less than 20% thickening of the diaphragm muscle during inspiration is diagnostic of diaphragmatic paralysis. Ultrasonography can also be used to serially monitor patients with diaphragmatic paralysis for recovery.

Phrenic nerve conduction studies can be carried out with placement of an oesophageal electrode to record diaphragmatic contractions and stimulation of the nerve in the neck either with surface stimulation or with a monopolar needle electrode at the level of the cricoid cartilage. Alternatively diaphragmatic electromyography may be carried out. The two tests are complementary. Electromyography may reveal a neuropathic versus myopathic pattern, depending on the etiology. This can be accomplished by stimulation of the phrenic nerve at the neck. Phrenic nerve stimulation can be done with electrical (surface or needle electrodes) and magnetic stimulation. Operator expertise is an important factor in testing. Technical issues with electromyography include proper electrode placement to avoid "cross-talk" from adjacent muscles and variable results due to variable subcutaneous fat among individuals. Using intraesophageal EMG electrodes is an alternative technique to avoid these issues. A method of unilateral magnetic stimulation of the phrenic nerve with concurrent assessment of diaphragm EMG and transdiaphragmatic pressures has also been described.

Measuring the vital capacity in the upright and supine positions is the most important part of the pulmonary function test. Diaphragmatic paralysis reduces the measured compliance of the lungs and a restrictive pattern can develop. Normally, vital capacity in recumbency decreases by 10%. In contrast, patients with unilateral diaphragmatic paralysis show a 15-30% decrease in vital capacity in supine position. This decrease is from cephalad displacement of abdominal contents.Pulmonary function test results, however, are not always consistent and do not always correlate with the severity of dyspnea from diaphragmatic paralysis.

Patients with diaphragmatic dysfunction and paralysis have a decrease in maximal inspiratory pressures (Pi,max). These patients cannot generate high negative inspiratory pressures. Therefore, the Pi,max in these patients is often reduced relative to normal values (Pi,max <70% predicted). Important to note is that decreased maximal pressures are the hallmark of diaphragmatic paralysis.

The transdiaphragmatic pressure is the criterion standard for diagnosis. Normal transdiaphragmatic pressure is approximately 148 cm water in men and 122 cm water in women. Unilateral diaphragmatic paralysis is associated with a maximal transdiaphragmatic pressure of greater than 70 cm water, and thus does not significantly effect transdiaphragmatic pressure generation during normal ventilatory behaviors, but can compromise higher-force, nonventilatory, behaviors like coughing or sneezing and also exercise breathing. Twitch transdiaphragmatic pressures after bilateral magnetic phrenic nerve stimulation are frequently used as a non-volitional assessment to confirm the presence of diaphragm weakness.

The functional limitations in individuals with respiratory disorders are not exclusively related to dyspnea. For example, balance impairments and resulting risk of falling are increasingly recognized issues in patients with COPD. Regarding the fact that postural balance is especially impaired in COPD patients with inspiratory muscle weakness, it can be hypothesized that diaphragm dysfunction plays an important role in the observed balance impairments. This is supported by the fact that the diaphragm is not only the principal inspiratory muscle, but also plays an important role in stabilizing the trunk during balance tasks. However, it remains unknown whether patients with diaphragm paresis show balance impairments, and whether these can be attributed to a dysfunction of the diaphragm. Furthermore, Kaufman et al. who followed up 180 patients with diaphragmatic paralysis, suggested that also low back pain might be associated with this disorder due to the fact that the postural function of the diaphragm is often disturbed in patients with low back pain. Also, individuals with low back pain show an increased diaphragm fatigability. However, neither the relation between diaphragmatic paralysis and postural control, neither between diaphragmatic paralysis and low back pain has been investigated yet.

Treatment options for UDP are limited. Diaphragmatic plication via mini thoracotomy is sometimes considered in the University Hospital Leuven if severe symptoms persist for longer than 12 months after initial diagnosis. Preliminary data indicate that daily inspiratory muscle strength and endurance training can lead to increased nondiaphragmatic inspiratory muscle recruitment and help those with symptoms from diaphragmatic paralysis. Randomized controlled trials comparing intervention groups with improvements achieved by natural recovery in the first months after diagnosis are however so far lacking. In addition there is a lack of comparable data between healthy subjects and patients.

The objective of the current study is therefore to investigate the effects of daily inspiratory muscle training in the first 6 months following diagnosis of unilateral diaphragmatic paralysis. A second objective is to compare (changes in) respiratory muscle function and activation patterns between healthy control subjects and patients. The investigators hypothesize that respiratory muscle training in symptomatic patients with UDP (in comparison with a control group) will reduce symptoms of exertional dyspnea (primary outcome) and will improve respiratory muscle function (at rest and during exercise) and pulmonary function (sitting and supine). Secondly, we hypothesize that the (changes in) recruiting patterns of diaphragmatic and non-diaphragmatic muscles will differ between healthy control subjects and patients both at baseline and in response to the intervention.

2. SPECIFIC OBJECTIVES

1. Investigate effects of IMT on intensity and quality of dyspnea perception in symptomatic patients with unilateral diaphragm paralysis during exercise
2. To identify and distinguish mechanisms responsible for dyspnea reduction after the intervention by exploring inter-relationships between the post-intervention change in dyspnea and changes in relevant measures of respiratory muscle function at rest and during exercise.
3. To compare changes in respiratory muscle recruitment patterns and respiratory neural drive to the diaphragm, as well as scalene, sternocleidomastoid and parasternal intercostal muscles in response to 6 months of inspiratory muscle strength- or endurance training during exercise.
4. To compare differences in (changes in) respiratory muscle recruitment patterns and respiratory neural drive to the diaphragm, as well as scalene, sternocleidomastoid and parasternal intercostal muscles, and postural control between healthy controls and patients.

ELIGIBILITY:
Inclusion Criteria for UDP patients:

* Stable, symptomatic adult UDP patients (age ≥18 yrs)
* UDP due to presumed neuralgic amyotrophy
* UDP after surgery/anesthesia (as long as there is no trauma/complete section of the phrenic nerves)
* idiopathic UDP
* UDP patients with Baseline Dyspnea Index (BDI) equal or lower than 9 out of 12.
* UDP patients who have reduced Pi,max (<70% of predicted normal value), reduced vital capacity (<75% predicted normal value in sitting and more than 15% reduction when performed supine compared to sitting).

Exclusion Criteria for UDP patients:

* underlying cardiac or respiratory disease that explains symptoms of dyspnea
* malignancy (i.e. metastatic lung cancer)
* diagnosed psychiatric or cognitive disorders
* concomitant progressive neurological, neuromuscular, or vestibular disorders
* severe orthopedic problems that have a major impact on performance of functional tests

Healthy adult (age ≥18 yrs) control subjects:

- recruitement via two methods. First, friends and family of the MSc student involved in this project will be asked to participate. Secondly, posters with information about the study will be displayed in the University hospital Leuven.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Dyspnea BORG category ratio 10 scale (scores from 1 to 10; higher score = worse outcome = more dyspnea) | pre-post 6 months intervention
  Difference in dyspnea intensity perception on a 10-point Borg scale at comparable time points during constant work rate cycling exercise pre-post intervention between groups.

SECONDARY OUTCOMES:
Respiratory muscle function | pre-post 6 months intervention and during every supervised IMT session in the hospital
  Pi,max will be recorded using the technique proposed by Black and Hyatt. Pes,max, Pgas,max, and Pdi,max values will be obtained during maximal sniff and cough maneuvers.Twitch Pdi will also be measured after uni- and bilateral magnetic phrenic nerve stimulation. Inspiratory muscle endurance will be tested with a protocol that we have recently established.
Phrenic nerve conduction | pre-post 6 months intervention
  Magnetic stimulation of the phrenic nerve in the neck in combination with diaphragmatic surface electromyography will be carried out to characterize phrenic nerve conduction.
Maximal end endurance exercise capacity | pre-post 6 months intervention
  A constant work rate (CWR) cycling test will be performed at 75% of the peak work rate achieved during a maximal incremental cardiopulmonary exercise test (CPET) to assess all main outcomes. CPET will be conducted on an electronically-braked cycle ergometer (Ergoline 800s; SensorMedics, Yorba Linda, CA) with detailed metabolic and cardiopulmonary measurements (SensorMedics Vs229d). On visit three (following IMT) two CWR tests will be performed. One until symptom limitation (tlim) and another until tlim of visit 2 to assess locomotor muscle fatigue at isotime as previously described by Amann et al. Subjects will rate intensity of breathing discomfort (dyspnea), unpleasantness of breathing, breathing-related anxiety, and leg discomfort, using the modified 10-point Borg scale. Qualitative descriptors of dyspnea will be collected at end-exercise.
Respiratory effort and neural respiratory drive to the diaphragm | pre-post 6 months intervention
  Pes, Pgas, Pdi and diaphragm electromyography (EMGdi) will be recorded continuously during cycle exercise using a multipair esophageal electrode catheter system. Surface EMG recordings of scalene and intercostal muscles will be performed according to a technique described by Duiverman et al.
Neural respiratory drive to breathing muscles | pre-post 6 months intervention
  Surface EMG recordings of scalene and intercostal muscles will be performed according to a technique described by Duiverman et al.
Pulmonary function (sitting and supine position) | pre-post 6 months intervention and during every supervised IMT session in the hospital
  Spirometry and whole body plethysmography will be performed according to the European Respiratory Society guidelines for pulmonary function testing (Vs62j body plethysmograph, SensorMedics, Yorba Linda, CA). (Quanjer PH, Tammeling GJ, Cotes JE, et al. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl 1993;16:5-40.) Changes in FEV1 (L), FVC (L), FRC (L) and RV (L) will be registered.
Severity of dyspnea pre intervention | pre-post 6 months intervention
  Assessed with Baseline throughout three categories: functional impairment, magnitude of task and magnitude of effort. A patient is asked open-ended questions regarding the symptoms. Following specific criteria, the observer is able to grade the degree of impairment (ranged 0-4) related to dyspnea for all three components. The range for the total score is 0-12. Lower score indicates a worse outcome.
Change in Severity of dyspnea post intervention | pre-post 6 months intervention
  Assessed with Transition Dyspnea Index (TDI) to assess changes over time. Patients report a slight, moderate or marked change, worse or better in comparison with BDI. A sum of the scores ranges between -9 and +9 where 0 indicates no change compared to baseline, a higher positive result indicates worsening of the condition and a lower negative result bigger improvement.
Dyspnea during daily life | pre-post 6 months of intervention
  Clinical grade of breathlessness is assessed on 5 point (1 to 5) Medical Research Council Dyspnea Scale. Higher score means more dyspnea and a worse outcome.
Postural control | pre-post 6 months intervention
  The participants will be asked to stand upright on a force plate. Displacements of the center of pressure (CoP) in anterior-posterior direction will be estimated from raw force plate data using the equation: CoP = Mx/Fz. Root mean square values of the CoP displacements will be used for the analysis of postural stability measures
Low back pain | pre-post 6 months intervention
  Disability related to low back pain will be evaluated using the Oswestry Disability Index, version 2 (adapted Dutch version) (ODI-2). A patient scores the impact of LBP on his functional ability in 10 domains of activities in daily life where each domain or item consists of 6 statements (scored 0-5). The total score is a sum ranging from 0 to 100 where higher score indicates a worse outcome (i.e. higher disability).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium